CLINICAL TRIAL: NCT07292623
Title: Effects of Transcutaneous Stimulation of the Auricular Branch of the Vagus Nerve in Older Adults
Brief Title: Effects of Transcutaneous Vagus Nerve Stimulation in Older Adults
Acronym: tVNS_older
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Alicia Martínez Rodríguez, Lecturer; Faculty of Physical Therapy. Researcher; Psychosocial Intervention and Functional Rehabilitation Group, Universidade da Coruña
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/295_I
Record Dates: First submitted 2025-11-29; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Older Adults Without Any Specific Clinical Condition; Autonomic Nervous System Imbalance; Transcutaneous Vagus Nerve Stimulation
Keywords: Transcutaneous Electric Nerve Stimulation; Vagus Nerve; Ear Auricle; Heart Rate; Aged; Voice; Saliva; Postural Balance; Tremor; Executive Function
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Intervention Model Description: All participants will undergo both conditions, placebo and real location, in a randomly assigned order. Placebo stimulation will be performed in a different location, using the same electrical parameters. The second session will be performed in the same way, but using the application not used in the previous session (placebo or active, as appropriate).
  Each session will follow this order:
  10 minutes (min) of acclimatization, connection of equipment and checking that the chest band is working; 10 to 35 min performance of the first set of tests; from 35 to 40 min measurement of heart rate variability (HRV); 40-45 min, searching for the highest intensity tolerated without discomfort- initiation of transcutaneous vagus nerve stimulation (sham or active tVNS); 45-50 min, HRV; from 50 to 75´ new performance of the set of tests with tVNS; 75-80 min final HRV; 80 min- tolerance, adverse effects (and 48 h after), blinding
Who Masked: Participant, Investigator
Masking Description: The volunteers will be randomized by sex to begin with one of two electrode locations: cymba concha and cavum concha at the left ear (active session); or scapha and lobule at the left ear (sham-session). These two interventions will be denominated as Transcutaneous Vagus Electrical Nerve Stimulation (t-VNS) and Sham Transcutaneous Vagus Electrical Nerve Stimulation (sham t-VNS). Allocation concealment, stratified by sex, will be ensured as the person will choose a piece of paper with the assignment coded with numbers (real/placebo) from a bag containing all the coded options that only the person applying the stimulation will see and understand (coded). The researcher analysing the results does not know whether condition 1 or 2 corresponds to the placebo or active location.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tVNS (Active Comparator): While acclimatization of the participant (10 minutes) the different tests will be explained, the chest strap will be placed, its synchronization with the HRV measurement system will be checked, and the TENS equipment will be placed on the waist using a fanny pack.
  The pre-stimulation assessment will be carried out (from 10 to 40 minutes after initiating the session). Participants will be allowed to try each one to familiarize themselves with it. All the tests will be performed (tremor, saliva, Flanker, balance, voice, Heart Rate Variability- HRV). At the end of this first part, the stimulation will be applied at the left ear in the area innervated by the vagus nerve (concha and cymba concha),and all the variables will be measured again in the same order during the actual electrical stimulation, after a new HRV measurement (from 45 to 75´). Then, the last HRV measurement will be taken and the participant will be asked about tolerance, the occurrence of adverse effects, and blinding.
  Interventions: Device: Active location tVNS
- Sham tVNS (Sham Comparator): At the beginning, the different tests will be explained, the chest strap will be placed, its synchronization with the HRV measurement system will be checked, and the TENS equipment will be placed on the waist using a fanny pack.
  Next, the pre-stimulation assessment will be carried out. Participants will be allowed to try each one to familiarize themselves with it. All the tests will be performed (tremor, saliva, Flanker, balance, voice, Heart Rate Variability- HRV). At the end of this first part, the stimulation will be applied at the left ear in the area not innervated by the vagus nerve (scapha) and all the variables will be measured in the same order during the sham electrical stimulation, after a new HRV measurement. Then, the last HRV measurement will be taken and the participant will be asked about tolerance, the occurrence of adverse effects, and blinding.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Active location tVNS — The tVNS will be performed at 20 Hz and 200 microseconds, in the area innervated by the auricular branch of the vagus nerve (cymba concha and concha) in the active location.
  The intensity will be set above the sensory threshold (intense tingling sensation) but below the level of discomfort. The TENS will be set to 27 seconds of working time, with a 3-second ramp-up and 90 seconds off. It will last until the end of the last HRV test.
  Other Names: tVNS; aVNS; auricular vagus nerve stimulation; Active tVNS
  Arms: Active tVNS
Device: Sham Comparator — The tVNS will be performed at 20 Hz and 200 microseconds, in the area not innervated by by the auricular branch of the vagus nerve (scapha) for sham TENS.
  The intensity will be set above the sensory threshold (intense tingling sensation) but below the level of discomfort. The TENS will be set to 27 seconds of working time, with a 3-second ramp-up and 90 seconds off. It will last until the end of the last HRV test.
  Other Names: Sham tVNS; sham aVNS; Sham auricular vagus nerve stimulation
  Arms: Sham tVNS

SUMMARY:
The autonomic nervous system consists of two branches, the sympathetic and the parasympathetic, which must work in balance. Its functioning can be measured indirectly by heart rate variability, which is the time between heartbeats, which is not constant. The more it varies, the greater the role of the parasympathetic branch, and vice versa. However, with age, an imbalance can occur and the parasympathetic branch can play a lesser role, resulting in less heart rate variability (the times between heartbeats become more similar).

The aim of this study is to know if electrical stimulation in the ear can improve the balance between the two branches of the autonomic nervous system in older adults, comparing two different locations of application. The main questions to answer are:

Does applying electrical stimulation to a specific area of the ear improve the balance of the autonomic nervous system? Does it also help improve hand tremors, balance, concentration, saliva production, and voice quality?

DETAILED DESCRIPTION:
Electrical stimulation (ES) of the nervous system, also denominated as neuromodulation, has been investigated for diverse conditions as cardiovascular diseases, chronic pain and psychiatric conditions. It is unknown which locations and parameters can be more effective and better tolerated. The transcutaneous ES is a non-invasive technique which has fewer side-effects than subcutaneous vagus nerve stimulation.

The aim of this study is to analyze the acute effects of transcutaneous ES on autonomic nervous modulation by heart rate variability (HRV) and heart frequency (HF) in older adults who perceive themselves as healthy, comparing two different locations for the ES, before and after a battery of motor, cognitive and other tests.. In addition, the tolerance to the current and the side-effects will be compared.

Once the participants have given their informed consent and had been checked for exclusion criteria, are invited to an experimental session. Subjects will be advised to refrain from caffeine or alcohol for 12 h and vigorous exercise for at least 24h prior to the intervention. The volunteers will be randomized by sex to begin with one of two electrode locations: cymba concha and cavum concha at the left ear (active session); or scapha and lobule at the left ear (sham-session). These two interventions will be denominated as Transcutaneous Vagus Electrical Nerve Stimulation (t-VNS) and Sham Transcutaneous Vagus Electrical Nerve Stimulation (sham t-VNS). Allocation concealment, stratified by sex, will be ensured as the person will choose a piece of paper with the assignment coded with numbers (real/placebo) from a bag containing all the coded options that only the person applying the stimulation will see and understand (coded) The stimulation location will be wiped down with alcohol and the minimum intensity, at which the stimulus is perceived, will be registered. Subsequently, the intensity will be increased until reaching the discomfort threshold, and then decreased to a strong but well-tolerated sensation.

At the beginning of the intervention, the different tests will be explained to the participant, the chest strap will be placed, its synchronisation with the HRV measurement system will be checked, and the TENS equipment will be placed on the waist using a belt.

After 10 minutes, the pre-stimulation assessment will be carried out. At the beginning of each session, participants will be allowed to try each one to familiarise themselves with it. At the end of the session, the stimulation will be applied and the variables will be measured in the same order during the actual electrical stimulation or placebo, as appropriate.

The second session will be performed in the same way, but using the application not used in the previous session (placebo or active, as appropriate).

The participants will be asked upon completion of the session their presumed group assignment.

Adverse effects will be checked at the end of each session, and again 48 h after.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers aged 65 to 80, with BMI from 18.5 to less than 30, who consider themselves healthy and are able to maintain their balance for at least 1 minute without assistance, living in A Coruña (Spain), with a 50% allocation to each sex

Exclusion Criteria:

* systolic blood pressure above 160 mm Hg and diastolic blood pressure above 100 mm Hg,
* previous vagotomy, history of syncope in the last two years, or lack of reliable reading in heart rate variability
* presence of chronic pain (migraine, back, neck, shoulder, etc.) or being diagnosed with or receiving treatment for malignant, cardiovascular disease (excluding hyperlipidaemia and hypercholesterolaemia), respiratory, neurological or autonomic, metabolic (e.g. diabetes), osteoarticular of autoimmune origin (e.g. arthritis), psychiatric or history of treatment with antidepressants or anxiolytics
* impaired cognitive level
* presence of any contraindication or difficulty in applying TENS: pacemaker, defibrillator or any implanted electronic device, apprehension of electric current, burns or irritated skin or allergic reaction or any alteration in the area that prevents the electrode from being placed on the left ear;
* previous application of electrical stimulation to the ear

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
HRV | Change from pre-tVNS (baseline= post initial battery of tests, about minute 35 after initiating the session) and during tVNS (post second battery of tests, 5 minutes before the end of the session, about minute 70)
  Heart Rate Variability (HRV) using Kubios app and H10 polar heart rate monitor chest strap, in periods of 5 minutes:
  * Frequency domain; ratio LF/HF power will be calculated along with normalised LF/HF where baseline values will set to 1; Low frequency (LF, referred to HRV frequency band 0.04-0.15 Hz); High frequency (HF = HRV frequency band 0.15-0.4 Hz); absolute powers of LF, and HF bands (ms2); normalized power (powers of LF and HF bands in normalised units, %)
  * Time domain: RR (mean values of RR intervals in ms) ; SDNN (Standard deviation of RR intervals); RMSSD (Root mean square of successive RR interval differences, in ms)
  * Non-linear methods: the poincaré plot short term variability (SD1, ms); the poincaré plot long term variability (SD2, ms).
  * Global measures: Stress Index (SI), square root of Baevsky's stress index; Parasympathetic nervous system (PNS) index

SECONDARY OUTCOMES:
HRV | Change from pre-tVNS (baseline = post initial battery of tests, about minute 35 after initiating the session) and initial tVNS (5 minutes after setting the intensity of tVNS, about 45 minutes after initiating the session)
  Heart Rate Variability (HRV) using Kubios app and H10 polar heart rate monitor chest strap in periods of 5 minutes:
  * Frequency domain; ratio LF/HF power will be calculated along with normalised LF/HF where baseline values will set to 1; Low frequency (LF, referred to HRV frequency band 0.04-0.15 Hz); High frequency (HF = HRV frequency band 0.15-0.4 Hz); absolute powers of LF, and HF bands (ms2); normalized power (powers of LF and HF bands in normalised units, %)
  * Time domain: RR (mean values of RR intervals in ms) ; SDNN (Standard deviation of RR intervals); RMSSD (Root mean square of successive RR interval differences, in ms)
  * Non-linear methods: the poincaré plot short term variability (SD1, ms); the poincaré plot long term variability (SD2, ms).
  * Global measures: Stress Index (SI), square root of Baevsky's stress index; Parasympathetic nervous system (PNS) index; Sympathetic nervous system (SNS) index
  * Mean heart rate (beats/min)
  * ECG derived respiration (breaths/min)
Hand tremor | Change from pre-tVNS (baseline= initial battery of tests, about minute 10 to 15 after initiating the session) and during tVNS (post = second battery of tests, about 50 to 55 minutes after after setting the intensity of tVNS)
  The tremor in both hands will be measured with the app (G-Sensor Logger) for a minute, using a mobile phone secured to each hand (both hands)
Salive | Change from pre-tVNS (baseline= initial battery of tests, from minute 15 to 20 after initiating the session) and during tVNS (post second battery of tests, about 55 to 60 minutes after after setting the intensity of tVNS)
  To measure salivation, a dry cloth will be placed in the mouth and weighed after 2 minutes without swallowing to estimate the volume of saliva produced.
Flanker test | Change from pre-tVNS (baseline= initial battery of tests, about 20 minutes after initiating the session) and during tVNS (post second battery of tests = 60 minutes after initiating the session)
  The Flanker test is designed to assess selective attention and inhibitory function, deciding the direction of a central row, flanked by nontarget stimuli, which can be congruent (matching the target) or incongruent (opposite to the target). It will be done with both arms.
Balance test | Change from pre-tVNS (baseline= post initial battery of tests, from minute 25) and during tVNS (post second battery of tests = from minute 65)
  For balance, a baropodometric platform will be used and the centre of pressure area (mm), the ellipse area (mm2), the speed (mm/s)and the displacements in the axes of space (mm) will be measured, with eyes open and eyes closed, twice on each occasion
Voice | Change from pre-tVNS (baseline= post initial battery of tests, from minute 35) and during tVNS (post second battery of tests = from minute 75 after initiating the session)
  The PRAAT software will be used to test the voice twice, when sustaining till 10 seconds the vowel "a" and when reading a text at their usual volume. The intensity, the fundamental frequency (F0), the jitter and shimmer parameters and the HNR (Harmonic to Noise Ratio) will be measured
Tolerance | Immediately after the intervention (around the 80th minute after the start of the session)
  The level of tolerance of the entire stimulation (by electrical stimulation, by electrodes, or by both) will be measured on a VAS scale from 0 (no discomfort at all) to 10 (the discomfort would have prevented me from finishing the session)
Adverse effects | Immediately after the intervention, and after 48 hours of ending it
  A questionnaire will be used to test the presence, severity, persistence and causality of ear pain, headache, tingling, itching, redness, irritation, pressure, dizziness, nausea, vertigo, fatigue, vertigo, palpitations, tinnitus, unpleasant feeling, other

OTHER OUTCOMES:
Efficacy of sham intervention | Immediately after the intervention
  Participants will be asked what stimulation they think they have just received, active or placebo (or what is their best guess) and why.
Amplitude of electrical stimulation | When initiating tVNS or sham-located tVNS, that means, 40 minutes after the initiation of the session
  mA at the initial sensation of the current and mA used during the electrical stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Martínez-Rodríguez, Lecturer, Principal Investigator — Universidade da Coruña (University of A Coruna); Olalla Bello, Lecturer, Principal Investigator — Universidade da Coruña (University of A Coruna)
Locations (1):
- Faculty of Physiotherapy, A Coruña, La Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
The IPD that underlie results included in the publication will be shared in Zenodo, with a description of the codes and needed information to understand it
Supporting Information: SAP, CSR
Time Frame: Beginning 1 year after publication and with no ending while Zenodo will keep the data
Access Criteria: The results will be included in a document which will be shared by Zenodo to all the investigators interested in them by direct access.